CLINICAL TRIAL: NCT02210546
Title: A Multicenter Randomised Trial of Contrast-enhanced MR Imaging as a Breast Cancer Screening Tool Alternative to Mammography and Ultrasonography in Women at Intermediate Risk. Feasibility, and Short Term Results.
Brief Title: Contrast-enhanced MR Imaging as a Breast Cancer Screening in Women at Intermediate Risk
Acronym: MRIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Paolo Bruzzi (Other)
Responsible Party: Sponsor-Investigator, Prof. Paolo Bruzzi, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Organization: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RF-2009-1539582
Record Dates: First submitted 2013-05-27; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; intermediate risk
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnetic Resonance Imaging (MRI) (Experimental): Patients will undergo MRI yearly
  Interventions: Other: Magnetic Resonance Imaging (MRI)
- Mammography (Mx) + ultrasonography (US) (Other): Patients will undergo yearly two-view (Mx) and breast US
  Interventions: Other: Mammography (Mx) + ultrasonography (US)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI)
  Arms: Magnetic Resonance Imaging (MRI)
Other: Mammography (Mx) + ultrasonography (US)
  Arms: Mammography (Mx) + ultrasonography (US)

SUMMARY:
A multicenter randomized controlled trial to evaluate the performance of MRI, in terms of sensitivity, specificity, and predictive value, in the screening of women at intermediate risk of breast cancer.

Two surveillance programs will be compared. Women will be randomly assigned with a 1:1 ratio to:

1. Yearly two-view mammography (Mx) and breast ultrasonography (US) or
2. Yearly MRI.

DETAILED DESCRIPTION:
Women, who, due to an increased risk of invasive breast cancer, are offered a specific surveillance program, as a supplement to the standard screening activities which in Italy are based on mammography every two years starting at age 50.Women will be randomly assigned to Yearly two-view mammography (Mx) and breast ultrasonography (US) or to Yearly MRI.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-59 years with
* cumulative risk at 10 years of at least 5%, or a lifetime cumulative breast cancer risk ranging between 15% and 30% (equivalent to a relative risk of 2-6 as compared to a low risk woman of the same age). The lifetime cumulative risk of breast cancer will be computed using the IBIS Breast Cancer Risk Evaluation Tool (http://www.ems-trials.org/riskevaluator/); or mammographic density involving more than 75% of the breast area, based on the most recent mammogram. The evaluation of the composition of the mammary gland will be performed using the BI-RADS classification. Women with mammography in class 4 (i.e., >75% of glandular component) will be eligible for randomization.
* Written Informed consent

Exclusion Criteria:

* Signs or symptoms of breast cancer at enrolment;
* Previous diagnosis of ductal carcinoma in situ or invasive breast cancer;
* BRCA or p53 mutation carrier status;
* General contraindications to MRI (e.g. cardiac pacemaker, metal implants or history of severe allergic reaction after administration of contrast agent;
* Contraindications to any intravenous administration of contrast agent;
* Ongoing or planned pregnancy (for the duration of the study);
* Hormonal enhancement of ovarian function for assisted reproduction in the previous 3 years
* Presence of breast implants;
* Previous diagnosis of cancer at any site;
* Life-threatening diseases;
* Mental disability precluding informed consent to participate

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Rate of in situ and invasive breast cancers detected in the two arms of the study | 36 months
  The performance of MRI will be evaluated , in terms of sensitivity, specificity, and predictive value, in the screening of women at intermediate risk of breast cancer

SECONDARY OUTCOMES:
Number of patients per each clinical and pathological stage of invasive cancer detected in the two arms of the study | 3 years
Proportion of the different histological characteristics of cancers detected in the two arms | 3 years
Number of invasive diagnostic procedures in the two study arms. | 3 years
Number of interval cancers in the two study arms. | 3 years
Rate of eligible women who accept to enter the study. | 3 years
Compliance to the intervention in the two study arms. | 3 years
Average and interquartile range of the risk profiles computed according to IBIS Breast Cancer Risk Evaluation Tool in the two arms | 3 years
Number of cancers (in situ and invasive) detected in excess in the experimental arm compared to the conventional arm (overdiagnosis) after 10 years of follow up | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Petrillo, MD, Principal Investigator — Istituto Nazionale dei Tumori IRCCS Fondazione Pascale (Naples); Paolo Belli, MD, Principal Investigator — Policlinico Gemelli (Rome); Alessandro Del Maschio, MD, Principal Investigator — Ospedale san Raffaele (Milan); Laura Martincich, MD, Principal Investigator — IRCCS Candiolo (Turin); Massimo Bazzocchi, MD, Principal Investigator — AOU S.Maria della Misericordia (Udine); Piero Panizza, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori (Milan); Stefania Montemezzi, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; Federica Pediconi, MD, Principal Investigator — Azienda Policlinico Umberto I (Rome); Stefano Corcione, MD, Principal Investigator — Azienda Ospedaliero Universitaria (Ferrara); Massimo Calabrese, MD, Principal Investigator — IRCCS AOU S. Martino-IST (Genoa); Francesco Sardanelli, MD, Principal Investigator — IRCCS San Donato (Milan)
Locations (1):
- IRCCS Azienda Ospedaliera Universitaria S.Martino IST, Genova, Italy